CLINICAL TRIAL: NCT02592850
Title: Osteopathic Manipulative Treatment in Frequent Episodic Tension-type Headache: the EBOTTH Multicentric Study
Brief Title: Evidence-Based Osteopathy for Tension-Type Headache (EBOTTH)
Acronym: EBOTTH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems for satellite centers in obtaining ethical clearance.
Sponsor: University of Milano Bicocca (Other)
Collaborators: Italian School of Osteopathy and Manual Therapies (Other); Alpha Search Milano (Unknown)
Responsible Party: Principal Investigator, Tremolizzo Lucio, Assistant Professor of Neurology, University of Milano Bicocca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EBOTTH-1; 203 (Registry Identifier: UNIMIB Ethic Commettee)
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Tension-Type Headache
Keywords: Osteopathic manipulative treatment; Frequent Episodic Tension-Type Headache; Randomized Controlled Trial
MeSH Terms: conditions — Tension-Type Headache | interventions — Manipulation, Osteopathic; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental): Active manipulative treatment.
  Interventions: Other: osteopathic manipulative treatment
- Sham Osteopathic Manipulative Treatment (Sham Comparator): Sham manipulative treatment.
  Interventions: Other: sham

INTERVENTIONS:
Other: osteopathic manipulative treatment — This intervention will not be protocol-based but the treating D.O. will compulsory have to include the evaluation (and possible treatment) of temporo-mandibular joint disorders and cervical dysfunctions (semi-structured treatment). Specifically, OMT will focus on correcting those osteopathic dysfunctions found during the initial evaluation; both structural (including myofascial release and HVLA), visceral and craniosacral techniques will be administered as appropriate.
  Duration: 45 minutes. Administered once a week for four weeks.
  Other Names: OMT
  Arms: Osteopathic Manipulative Treatment
Other: sham — In this intervention, the operator will be restricted to the assessment of the cranial rhythmic impulse (CRI), temporo-mandibular joint disorders and cervical dysfunctions, spending a similar amount of time to that being spent on OMT-treated patients. Any found osteopathic dysfunction will not be corrected.
  Duration: 45 minutes. Administered once a week for four weeks.
  Other Names: SHAM-OMT
  Arms: Sham Osteopathic Manipulative Treatment

SUMMARY:
Tension-type headache (TTH) is a very common primary headache disorder, with important costs for both patients and society. Often these patients are not willing to take prophylactic medications and resort to complementary therapies. Osteopathic manipulative treatment (OMT) is an interesting option in such field, since it is characterized by a low profile of side effects.

In this study the investigators will assess the efficacy of OMT (semi-structured evaluation and "black box" treatment) in frequent Episodic TTH (ETTH) in an outpatient setting. Preliminary data for power calculation are already available (Rolle et al. 2014), and the investigators plan to recruit 264 ETHH patients by a multicentric, randomized, double-blind, sham-controlled design.

DETAILED DESCRIPTION:
Background:

Primary headache disorders are very common throughout the world, producing widespread and substantial disability and representing a concrete public-health priority. Tension-type headache (TTH) is the most common type of primary headache disorder, with a lifetime prevalence in the general population ranging between 30% and 78% in different studies. In general, headache is a chronic disorder with episodic manifestations that may range from few attacks/year up to daily episodes. Its impact on individuals' lives is greater than has generally been realized, including psychiatric, psychological and social correlates. The impact on patients can be very high, including ictal symptom burden, interictal burden, cumulative burden and impact on other people. The individual burden of TTH includes both symptoms occurring during the attacks (pain, eventually accompanied by no more than one of phonophobia or photophobia, according to International Classification of Headache Disorders) and elements of interictal burden, such as anxiety, mood disorders, affective distress and avoidance behavior. While present, symptoms may cause debility and prostration, and reduce functional ability. Even if patients with TTH generally are not unable to work, effectiveness and productivity may be consistently reduced. This secondary disability is quite significant because headache in general is most common in people between their teens and 50-60 years of age, the productive years. The elements of interictal burden, instead, may continuously affect wellbeing and impair quality of life. Moreover, TTH has a substantial impact on the health system, due to both direct and indirect financial cost. The high prevalence of TTH, considering its individual impact and huge financial costs, has important implications for health policy, since it is a source of high but potentially reducible socioeconomic burden. Essentially, TTH management is a public-health priority.

On the clinical side, tension-type headache has been defined as a multifactorial disorder, conceivably implying the need for tailored treatment strategies. Headache-related disability can usually be reduced by identifying and avoiding triggers combined with pharmacologic and non-pharmacologic treatment (such as relaxation and stress management techniques or physical therapies), but effective treatment modalities are still lacking. Particularly, symptomatic drugs are effective for episodes of TTH, whereas preventive treatment (indicated for frequent and chronic TTH) is, on average, barely effective, and do not display good tolerability. Patients are turning to complementary or alternative therapies for headaches, including osteopathic manipulative therapy (OMTh). One previous pilot study carried out by the investigators has suggested an efficacy for OMTh in frequent episodic TTH, that might represent an alternative treatment strategy to prophylactic drugs. Frequent episodic TTH (ETTH) was chosen for this study since it is the most common diagnostic category with indications for prophylactic drug management. To date there is no rigorously tested evidence that manual therapies in general have a positive effect on TTH, as many reviewers have found. Conflicting results in previous studies might be due both to the low number of clinical trials and an indiscriminate application of different techniques. Some studies, however, have demonstrated positive effects of manipulative therapy.

A systematic review found spinal manipulative therapy as effective as commonly used first-line prophylactic medications for both TTH and migraine headaches, but the Authors emphasized that their conclusions were based on only a few trials, raising the question of whether their analysis was methodologically adequate. A more recent systematic review concluded that spinal manipulation might alleviate TTH but that the small quantity of available data prevented any definitive conclusions. The combination of physical therapies with medications, can also increase the success of the treatment, particularly in case of comorbid mood disorders and unremitting headaches, as previously suggested. Although results of these and others published studies suggest positive effects, OMTh has rarely been rigorously tested for the care of patients with headache in general.

OMTh is not free of costs but is plausibly characterized by fewer contraindications and adverse events than conventional pharmacological treatments, and particularly indicated for patients not compliant with drug regimens and those at increased risk of adverse drug effects. Notably, there is disparity between patient perceptions and clinical definitions of adverse events, as a conceptual model with four inter-related components (expectation, personal investment, osteopathic encounter and clinical change) has suggested. Patients might report mild effects following OMTh and in general all forms of manual therapy, but these effects should not be strictly regarded as adverse events. Our previous pilot trial did not observe adverse events among ETTH patients belonging to both arms of the study (treatment and sham). Exceedingly rare serious adverse events may be observed after spine manipulation, only one of many different techniques usually administered in osteopathic clinical field and recommendations have been already published to meet the requirements of the principles of prevention and precaution. For example, minor unwanted effects of prior manipulation should be searched routinely and taken as contraindication for future spinal manipulations. Great care should be taken when particular anatomic conditions such as cord encroachment or increased vertebra-basilar risk are present. Certainly, besides effectiveness, still to be completely proven, the financial impact of OMTh on subjects and health systems could be also a topic of appraisal for future comparative studies.

However, considering all the exposed priorities in this field, the investigators decided to firstly address in a RCT the question of OMTh efficacy versus OMTh-sham treatment in ETTH.

Aims:

This is a protocol for a randomized controlled trial (RCT) exploring the efficacy of OMTh in ETTH with respect to OMTh-sham treatment by a single blinded multicenter design.

If OMTh effectiveness could be demonstrated in these patients, two putative repercussions in ETTH management might be expected: (a) increased compliance; (b) lower rate of side effects. Furthermore, OMTh would increase the range of available strategies for managing ETTH in clinical practice, perhaps even as an add-on therapy.

Study Design:

This is a multi-centre, double-blinded, randomized, sham-treatment (SHAM)-controlled study using an experimental design.

Presumed ETTH patients will be screened at pre-selected primary care settings (general practitioners), and the diagnosis of TTH reviewed (time -30, or T-30) by a neurologist that will ask patients to complete the headache diary for 30 days before randomization. Diaries will be reviewed at time 0 (T0; baseline) by a blind-rater D.O. that will decide if the number of attacks is compatible with the diagnosis of ETTH, allowing randomization. The blind-rater will perform an osteopathic structural examination that will compulsory include (semi-structured evaluation) also the assessment of temporo-mandibular joint disorders and cervical dysfunctions (TMJD and CD) in order to define putative goals of OMT that will be used for scoring a Goal Attainment Scale (GAS, see below Outcomes) without involving the treating D.O. that will operate independently. Furthermore, patients will be asked to complete the Headache Disability Inventory (HDI) and the Headache Impact Test-6 (HIT-6).

Randomization will be performed by the coordinating centre (Univ. of Milano-Bicocca, Italy) by randomly pre-generated lists; the coordinating centre, without informing the blind-rater, will communicate to the local Osteopathic Clinic these details. Patients will be given instructions to start treatment (OMT vs. SHAM in blind) that will be administered by a treating D.O. unblinded to treatment allocation. Patients will receive 4 weekly treatments completing the headache diary along the whole study (up to T120). The blind-rater will review diaries relative to the each previous period and ask patients to complete the HDI/HIT-6 at 30 days (T30, end of treatment), 60 days (T60, follow-up-1), 90 days (T90, follow-up-2) and 120 days (T120, end of study) with respect to randomization (T0). An osteopathic structural examination will be performed again at T120 (end of study) for GAS scoring. A central database will be filled.

Inclusion criteria will be: (1) a diagnosis of ETTH according to current International Headache Society guidelines; (2) willing to comply with the RCT procedures.

Exclusion criteria will be: (1) patients under 18 or over 65 years of age; (2) use during the previous three months of drugs for acute headache on ten or more days per month; (3) duration of disease less than one year; (4) history of major psychiatric diseases, significant cognitive disorders, significant chronic pain other than headache, or in general from a secondary headache; (5) any kind of ongoing prophylactic treatment or taking place during the whole study period; (6) estroprogestinic therapy started or modified during the whole study period.

Patients will be blindly allocated to (A) an experimental arm (OMT) and (B) a control arm (SHAM), i.e., manual perceptive technique without correction of any observed osteopathic disorder. In order to minimize the perceived differences, both groups will undergo to osteopathic structural examination, with a similar amount of time being spent on each session. OMT will not be protocol-based but the treating D.O. will compulsory have to include the evaluation (and possible treatment) of TMJD and CD (semi-structured treatment). Specifically, OMT will focus on correcting those osteopathic dysfunctions found during the initial evaluation; both structural (including myofascial release and HVLA), visceral and craniosacral techniques will be administered as appropriate. As regards the sham treatment, the operator will be restricted to the assessment of the cranial rhythmic impulse (CRI) in patients, spending a similar amount of time to that being spent on OMT-treated patients.

Primary outcome will be the change at T120 in patient-reported headache frequency of at least 30% with respect to the control group (based on the previous pilot study, Rolle et al. 2014). Secondary outcomes will include: (a) any significant reduction over time or with respect to the control group of the average headache intensity based on a scale between 0 (absence of pain) and 5 (worst perceived pain) (considered more sensible with respect to a 0-to-3 scale, see Rolle et al. 2014); (b) any significant reduction over time or with respect to the control group of the over-the-counter medication usage; (c) any significant reduction over time or with respect to the control group of the HDI/HIT-6 scores; (d) any significant reduction over time or with respect to the control group in patient-reported headache frequency. Tertiary outcome will be: any significant reduction over time or with respect to the control group of the blind-rater evaluation of the osteopathic effects of the whole treatment with respect to the attainments he initially proposed. This score will be assessed purely in terms of correction of those osteopathic dysfunctions that were detected at T0, by using the GAS, with a five-point score ranging from: -2 (much less than expected outcome), to -1 (less than expected outcome), to 0 (expected outcome reached), to +1 (greater than expected outcome), to +2 (much greater than expected outcome).

Finally, side effects will be recorded at each visit. Patients will be instructed to immediately report serious adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 and ≤65 years-old,
* diagnosis of frequent episodic tension-type headache according to the International Headache Society guidelines,
* frequency of attacks ≥3/month,
* willing to adhere to study procedures,
* signed informed consent

Exclusion Criteria:

* age <18 or >65 years-old,
* headache duration less than one year,
* history of: major psychiatric disorders, relevant cognitive deficits, chronic pain other than headache, secondary headaches,
* any type of headache prophylactic treatment ongoing or started during the study,
* hormonal therapy started or modified during the study,
* participating to other clinical trials,
* not willing to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Headache frequency | 4 months
  average reduction of headache frequency between the two arms and/or over time obtained from the headache diary (n/month)

SECONDARY OUTCOMES:
Headache intensity | 4 months
  average reduction of headache intensity between the two arms and/or over time obtained from the headache diary (average value; scale 0-5)
Symptomatic Drugs | 4 months
  average modification of symptomatic drug use between the two arms and/or over time obtained from the headache diary (n/month)
Headache Disability Inventory (HDI) | 4 months
  average modification of HDI scores between the two arms and/or over time
Headache Impact Test-6 (HIT-6) | 4 months
  average modification of HIT-6 scores between the two arms and/or over time
Side effects | 4 months
  any type of adverse event

OTHER OUTCOMES:
Goal Attainment Scale (GAS) for osteopathic dysfunction | 4 months
  any modification of any osteopathic dysfunction found at study entry between the two arms and/or over time (score between -2 and +2)

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Tremolizzo, MD, PhD, Principal Investigator — University of Milano-Bicocca, Italy; Guido Rolle, DO, MD, Study Director — Italian School of Osteopathy and Manual Therapies

REFERENCES:
- [Background] Stovner Lj, Hagen K, Jensen R, Katsarava Z, Lipton R, Scher A, Steiner T, Zwart JA. The global burden of headache: a documentation of headache prevalence and disability worldwide. Cephalalgia. 2007 Mar;27(3):193-210. doi: 10.1111/j.1468-2982.2007.01288.x. PMID 17381554
- [Background] Jensen R, Stovner LJ. Epidemiology and comorbidity of headache. Lancet Neurol. 2008 Apr;7(4):354-61. doi: 10.1016/S1474-4422(08)70062-0. PMID 18339350
- [Background] Schwartz BS, Stewart WF, Simon D, Lipton RB. Epidemiology of tension-type headache. JAMA. 1998 Feb 4;279(5):381-3. doi: 10.1001/jama.279.5.381. PMID 9459472
- [Background] Rasmussen BK, Jensen R, Schroll M, Olesen J. Epidemiology of headache in a general population--a prevalence study. J Clin Epidemiol. 1991;44(11):1147-57. doi: 10.1016/0895-4356(91)90147-2. PMID 1941010
- [Background] Stovner LJ, Zwart JA, Hagen K, Terwindt GM, Pascual J. Epidemiology of headache in Europe. Eur J Neurol. 2006 Apr;13(4):333-45. doi: 10.1111/j.1468-1331.2006.01184.x. PMID 16643310
- [Background] Stovner LJ, Hagen K. Prevalence, burden, and cost of headache disorders. Curr Opin Neurol. 2006 Jun;19(3):281-5. doi: 10.1097/01.wco.0000227039.16071.92. PMID 16702836
- [Background] Stovner LJ, Andree C. Prevalence of headache in Europe: a review for the Eurolight project. J Headache Pain. 2010 Aug;11(4):289-99. doi: 10.1007/s10194-010-0217-0. Epub 2010 May 16. PMID 20473702
- [Background] Jensen R. Diagnosis, epidemiology, and impact of tension-type headache. Curr Pain Headache Rep. 2003 Dec;7(6):455-9. doi: 10.1007/s11916-003-0061-x. PMID 14604504
- [Background] Holroyd KA, Stensland M, Lipchik GL, Hill KR, O'Donnell FS, Cordingley G. Psychosocial correlates and impact of chronic tension-type headaches. Headache. 2000 Jan;40(1):3-16. doi: 10.1046/j.1526-4610.2000.00001.x. PMID 10759896
- [Background] Beghi E, Bussone G, D'Amico D, Cortelli P, Cevoli S, Manzoni GC, Torelli P, Tonini MC, Allais G, De Simone R, D'Onofrio F, Genco S, Moschiano F, Beghi M, Salvi S. Headache, anxiety and depressive disorders: the HADAS study. J Headache Pain. 2010 Apr;11(2):141-50. doi: 10.1007/s10194-010-0187-2. Epub 2010 Jan 27. PMID 20108021
- [Background] Steiner TJ, Stovner LJ, Katsarava Z, Lainez JM, Lampl C, Lanteri-Minet M, Rastenyte D, Ruiz de la Torre E, Tassorelli C, Barre J, Andree C. The impact of headache in Europe: principal results of the Eurolight project. J Headache Pain. 2014 May 21;15(1):31. doi: 10.1186/1129-2377-15-31. PMID 24884549
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Lenaerts ME. Burden of tension-type headache. Curr Pain Headache Rep. 2006 Dec;10(6):459-62. doi: 10.1007/s11916-006-0078-z. PMID 17087872
- [Background] Linde M, Gustavsson A, Stovner LJ, Steiner TJ, Barre J, Katsarava Z, Lainez JM, Lampl C, Lanteri-Minet M, Rastenyte D, Ruiz de la Torre E, Tassorelli C, Andree C. The cost of headache disorders in Europe: the Eurolight project. Eur J Neurol. 2012 May;19(5):703-11. doi: 10.1111/j.1468-1331.2011.03612.x. Epub 2011 Dec 5. PMID 22136117
- [Background] Bendtsen L, Jensen R. Treating tension-type headache -- an expert opinion. Expert Opin Pharmacother. 2011 May;12(7):1099-109. doi: 10.1517/14656566.2011.548806. Epub 2011 Jan 20. PMID 21247362
- [Background] Bendtsen L, Jensen R. Tension-type headache. Neurol Clin. 2009 May;27(2):525-35. doi: 10.1016/j.ncl.2008.11.010. PMID 19289230
- [Background] Fumal A, Schoenen J. Tension-type headache: current research and clinical management. Lancet Neurol. 2008 Jan;7(1):70-83. doi: 10.1016/S1474-4422(07)70325-3. PMID 18093564
- [Background] Jensen R, Rasmussen BK. Burden of headache. Expert Rev Pharmacoecon Outcomes Res. 2004 Jun;4(3):353-9. doi: 10.1586/14737167.4.3.353. PMID 19807317
- [Background] Barbanti P, Egeo G, Aurilia C, Fofi L. Treatment of tension-type headache: from old myths to modern concepts. Neurol Sci. 2014 May;35 Suppl 1:17-21. doi: 10.1007/s10072-014-1735-3. PMID 24867829
- [Background] Mathew PG, Mathew T. Taking care of the challenging tension headache patient. Curr Pain Headache Rep. 2011 Dec;15(6):444-50. doi: 10.1007/s11916-011-0223-1. PMID 21845469
- [Background] Rolle G, Tremolizzo L, Somalvico F, Ferrarese C, Bressan LC. Pilot trial of osteopathic manipulative therapy for patients with frequent episodic tension-type headache. J Am Osteopath Assoc. 2014 Sep;114(9):678-85. doi: 10.7556/jaoa.2014.136. PMID 25170037
- [Background] Fernandez-de-Las-Penas C, Alonso-Blanco C, Cuadrado ML, Miangolarra JC, Barriga FJ, Pareja JA. Are manual therapies effective in reducing pain from tension-type headache?: a systematic review. Clin J Pain. 2006 Mar-Apr;22(3):278-85. doi: 10.1097/01.ajp.0000173017.64741.86. PMID 16514329
- [Background] Fernandez-de-las-Penas C, Alonso-Blanco C, San-Roman J, Miangolarra-Page JC. Methodological quality of randomized controlled trials of spinal manipulation and mobilization in tension-type headache, migraine, and cervicogenic headache. J Orthop Sports Phys Ther. 2006 Mar;36(3):160-9. doi: 10.2519/jospt.2006.36.3.160. PMID 16596892
- [Background] Tsao JC. Effectiveness of massage therapy for chronic, non-malignant pain: a review. Evid Based Complement Alternat Med. 2007 Jun;4(2):165-79. doi: 10.1093/ecam/nel109. Epub 2007 Feb 5. PMID 17549233
- [Background] Lenssinck MB, Damen L, Verhagen AP, Berger MY, Passchier J, Koes BW. The effectiveness of physiotherapy and manipulation in patients with tension-type headache: a systematic review. Pain. 2004 Dec;112(3):381-388. doi: 10.1016/j.pain.2004.09.026. PMID 15561394
- [Background] Astin JA, Ernst E. The effectiveness of spinal manipulation for the treatment of headache disorders: a systematic review of randomized clinical trials. Cephalalgia. 2002 Oct;22(8):617-23. doi: 10.1046/j.1468-2982.2002.00423.x. PMID 12383058
- [Background] Fernandez-de-Las-Penas C. Physical therapy and exercise in headache. Cephalalgia. 2008 Jul;28 Suppl 1:36-8. doi: 10.1111/j.1468-2982.2008.01618.x. PMID 18494995
- [Background] Jull G, Trott P, Potter H, Zito G, Niere K, Shirley D, Emberson J, Marschner I, Richardson C. A randomized controlled trial of exercise and manipulative therapy for cervicogenic headache. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1835-43; discussion 1843. doi: 10.1097/00007632-200209010-00004. PMID 12221344
- [Background] Torelli P, Jensen R, Olesen J. Physiotherapy for tension-type headache: a controlled study. Cephalalgia. 2004 Jan;24(1):29-36. doi: 10.1111/j.1468-2982.2004.00633.x. PMID 14687010
- [Background] Espi-Lopez GV, Rodriguez-Blanco C, Oliva-Pascual-Vaca A, Benitez-Martinez JC, Lluch E, Falla D. Effect of manual therapy techniques on headache disability in patients with tension-type headache. Randomized controlled trial. Eur J Phys Rehabil Med. 2014 Dec;50(6):641-7. Epub 2014 Apr 30. PMID 24785463
- [Background] Bronfort G, Assendelft WJ, Evans R, Haas M, Bouter L. Efficacy of spinal manipulation for chronic headache: a systematic review. J Manipulative Physiol Ther. 2001 Sep;24(7):457-66. PMID 11562654
- [Background] Posadzki P, Ernst E. Spinal manipulations for tension-type headaches: a systematic review of randomized controlled trials. Complement Ther Med. 2012 Aug;20(4):232-9. doi: 10.1016/j.ctim.2011.12.001. Epub 2011 Dec 29. PMID 22579436
- [Background] Sun-Edelstein C, Mauskop A. Complementary and alternative approaches to the treatment of tension-type headache. Curr Pain Headache Rep. 2008 Dec;12(6):447-50. doi: 10.1007/s11916-008-0076-4. PMID 18973739
- [Background] Hoyt WH, Shaffer F, Bard DA, Benesler JS, Blankenhorn GD, Gray JH, Hartman WT, Hughes LC. Osteopathic manipulation in the treatment of muscle-contraction headache. J Am Osteopath Assoc. 1979 Jan;78(5):322-5. No abstract available. PMID 581588
- [Background] Ajimsha MS. Effectiveness of direct vs indirect technique myofascial release in the management of tension-type headache. J Bodyw Mov Ther. 2011 Oct;15(4):431-5. doi: 10.1016/j.jbmt.2011.01.021. Epub 2011 Feb 11. PMID 21943616
- [Background] Voigt K, Liebnitzky J, Burmeister U, Sihvonen-Riemenschneider H, Beck M, Voigt R, Bergmann A. Efficacy of osteopathic manipulative treatment of female patients with migraine: results of a randomized controlled trial. J Altern Complement Med. 2011 Mar;17(3):225-30. doi: 10.1089/acm.2009.0673. Epub 2011 Mar 8. PMID 21385086
- [Background] Anderson RE, Seniscal C. A comparison of selected osteopathic treatment and relaxation for tension-type headaches. Headache. 2006 Sep;46(8):1273-80. doi: 10.1111/j.1526-4610.2006.00535.x. PMID 16942472
- [Background] Rajendran D, Bright P, Bettles S, Carnes D, Mullinger B. What puts the adverse in 'adverse events'? Patients' perceptions of post-treatment experiences in osteopathy--a qualitative study using focus groups. Man Ther. 2012 Aug;17(4):305-11. doi: 10.1016/j.math.2012.02.011. Epub 2012 Mar 15. PMID 22425134
- [Background] Tinel D, Bliznakova E, Juhel C, Gallien P, Brissot R. Vertebrobasilar ischemia after cervical spine manipulation: a case report. Ann Readapt Med Phys. 2008 Jun;51(5):403-14. doi: 10.1016/j.annrmp.2008.04.010. Epub 2008 May 28. English, French. PMID 18586346
- [Background] Cicconi M, Mangiulli T, Bolino G. Onset of complications following cervical manipulation due to malpractice in osteopathic treatment: a case report. Med Sci Law. 2014 Oct;54(4):230-3. doi: 10.1177/0025802413513451. Epub 2014 Jan 8. PMID 24402084
- [Background] Greenman PE, McPartland JM. Cranial findings and iatrogenesis from craniosacral manipulation in patients with traumatic brain syndrome. J Am Osteopath Assoc. 1995 Mar;95(3):182-8; 191-2. PMID 7751168
- [Background] Suh SI, Koh SB, Choi EJ, Kim BJ, Park MK, Park KW, Yoon JS, Lee DH. Intracranial hypotension induced by cervical spine chiropractic manipulation. Spine (Phila Pa 1976). 2005 Jun 15;30(12):E340-2. doi: 10.1097/01.brs.0000166511.59868.b7. PMID 15959358
- [Background] Hebert JJ, Stomski NJ, French SD, Rubinstein SM. Serious Adverse Events and Spinal Manipulative Therapy of the Low Back Region: A Systematic Review of Cases. J Manipulative Physiol Ther. 2015 Nov-Dec;38(9):677-691. doi: 10.1016/j.jmpt.2013.05.009. Epub 2013 Jun 17. PMID 23787298
- [Background] Noll DR, Degenhardt BF, Stuart M, McGovern R, Matteson M. Effectiveness of a sham protocol and adverse effects in a clinical trial of osteopathic manipulative treatment in nursing home patients. J Am Osteopath Assoc. 2004 Mar;104(3):107-13. No abstract available. PMID 15083985
- [Background] Vautravers P, Maigne JY. Cervical spine manipulation and the precautionary principle. Joint Bone Spine. 2000;67(4):272-6. PMID 10963073
- [Background] Vautravers P, Maigne JY. [Cervical spine manipulation: risks--benefit--assessment]. Rev Neurol (Paris). 2003 Nov;159(11):1064-6. French. PMID 14710030
- [Background] Murphy DR, Hurwitz EL, Gregory AA. Manipulation in the presence of cervical spinal cord compression: a case series. J Manipulative Physiol Ther. 2006 Mar-Apr;29(3):236-44. doi: 10.1016/j.jmpt.2006.01.001. PMID 16584950
- [Background] Cagnie B, Barbaix E, Vinck E, D'Herde K, Cambier D. A case of abnormal findings in the course of the vertebral artery associated with an ossified hyoid apparatus. A contraindication for manipulation of the cervical spine? J Manipulative Physiol Ther. 2005 Jun;28(5):346-51. doi: 10.1016/j.jmpt.2005.04.007. PMID 15965410